CLINICAL TRIAL: NCT03274219
Title: A Phase 1 Study of bb21217, an Anti-BCMA CAR T Cell Drug Product, in Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study of bb21217 in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 2seventy bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRB-402
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bb21217 Experimental Arm (Experimental)
  Interventions: Biological: bb21217

INTERVENTIONS:
Biological: bb21217 — autologous T cells transduced ex-vivo with anti-BCMA CAR lentiviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA, suspended in cryopreservative solution

SUMMARY:
Study CRB-402 is a 2-part, non-randomized, open label, multi-site Phase 1 study of bb21217 in adults with relapsed/refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
Part A of the study will be Dose Escalation followed by Part B, an expansion cohort.

Following consent, enrolled subjects will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (bb21217). Following manufacture of the drug product, subjects will receive lymphodepletion prior to bb21217 infusion. All subjects will then be followed for up to 60 months in Study CRB-402.

All subjects who complete the study, as well as those who withdraw from the study after receiving bb21217 for reasons other than death or meeting the early termination criteria, will be asked to continue to undergo long-term follow-up in a companion study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Diagnosis of MM with relapsed or refractory disease and have had at least 3 different prior lines of therapy with previous exposure to PI, IMiDs, and a CD38 antibody. Have undergone at least 2 consecutive cycles of treatment for each therapy, unless PD was the best response to the therapy. Refractory to their last line of therapy.
* Subjects must have measurable disease

Exclusion Criteria:

* Subjects with known central nervous system disease
* Inadequate hepatic function
* Inadequate renal function
* Inadequate bone marrow function
* Presence of active infection within 72 hours
* Subjects with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, recent significant traumatic injury, and other conditions
* Known human immunodeficiency virus (HIV) positivity
* Known hepatitis A virus (HAV), hepatitis B virus (HBV) or hepatitis C virus (HCV) positivity with evidence of ongoing infection.
* Pregnant or lactating women
* Previous history of an allogeneic bone marrow transplantation, treatment with any gene therapy based therapeutic for cancer, or BCMA-targeted therapy
* Inadequate pulmonary function defined as oxygen saturation (SaO2) <92% on room air
* Subjects who have a history of plasma cell leukemia, active plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS, or clinically significant amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), DLTs, and changes in laboratory results | Day 1 through Month 60
  Incidence of adverse events (AEs) and abnormal laboratory test results, including dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Disease-specific response criteria | Month 1 through Month 60
  • Disease-specific response criteria including, but not limited to: complete response (CR), very good partial response (VGPR), and partial response (PR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Anna Truppel-Hartmann, MD, Study Director — Genetix Biotherapeutics Inc.
Locations (11):
- United States (11):
  - UCSF Medical Center at Parnassus, San Francisco, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Insitute, Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- [Derived] Madduri D, Parekh S, Campbell TB, Neumann F, Petrocca F, Jagannath S. Anti-BCMA CAR T administration in a relapsed and refractory multiple myeloma patient after COVID-19 infection: a case report. J Med Case Rep. 2021 Feb 19;15(1):90. doi: 10.1186/s13256-020-02598-0. PMID 33608053